CLINICAL TRIAL: NCT06809530
Title: Intrathecal Administration of Dual Checkpoint Inhibitor in Combination With Pemetrexed in Patients With Leptomeningeal Metastasis: a Phase I/II Study
Brief Title: Intrathecal Dual Checkpoint Inhibitor (PD-1 and CTLA-4) in Combination With Pemetrexed for Leptomeningeal Metastasis
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Zhenyu Pan, Professor, Guangzhou Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IT-P-QL1706
Record Dates: First submitted 2025-01-26; First posted 2025-02-05 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-01

CONDITIONS: Leptomeningeal Metastasis; Pemetrexed; PD-1 Inhibitor; CTLA4; Solid Tumors
Keywords: Leptomeningeal metastasis; dual checkpoint inhibitor; pemetrexed
MeSH Terms: conditions — Meningeal Carcinomatosis | interventions — Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intrathecal Dual Checkpoint Inhibition in Combination with Pemetrexed (Experimental): This study is a prospective, single-arm, Phase I/II clinical trial. The primary objectives were to determine the recommended dose of intrathecal dual checkpoint inhibitor (PD-1 and CTLA-4, QL1706) in combination with pemetrexed and safety based on the incidence of treatment-related adverse events. Clinical response rate (CRR), progression-free survival related to leptomeningeal metastasis (LMPFS) and overall survival (OS) are also evaluated. Patients will have cerebrospinal fluid (CSF) and blood specimen collection for the evaluation of predictors (clinical, molecular, and/or immune) of the efficacy and safety of this regimen.
  Interventions: Drug: QL1706 (bispecific antibody targeting PD-1 and CLTA-4); Drug: Pemetrexed (Alimta)

INTERVENTIONS:
Drug: QL1706 (bispecific antibody targeting PD-1 and CLTA-4) — Intrathecal injection of PD-1/CTLA-4 bispecific antibody was administered every 2 weeks for 6 weeks during the induction phase, followed by monthly injections during the maintenance phase, until recurrence or death.
Drug: Pemetrexed (Alimta) — Pemetrexed (Alimta, Eli Lilly and Company) was administrated by intrathecal injection, first as induction therapy, twice per week for 2 weeks, followed by consolidation therapy, once per week for 4 weeks, then maintenance therapy, once per month until the patient's death, leptomeningeal metastasis progresses, or intolerable severe adverse events occurred.

SUMMARY:
This phase I/II study is to evaluate the recommended dose, safety, feasibility, and therapeutic response of intrathecal dual checkpoint inhibitor (targeting PD-1 and CTLA-4 with QL1706) in combination with pemetrexed in patients with leptomeningeal metastasis.

DETAILED DESCRIPTION:
This study is a prospective, single-arm, phase I/II clinical trial evaluating intrathecal dual checkpoint inhibitor (targeting PD-1 and CTLA-4 with the bispecific antibody QL1706) in combination with pemetrexed for the treatment of leptomeningeal metastasis.

Intrathecal pemetrexed is administered twice weekly for 2 weeks (induction phase), then weekly for 4 weeks (consolidation phase), and monthly thereafter (maintenance phase). Intrathecal QL1706 (a PD-1/CTLA-4 bispecific antibody) is given every two weeks during the six-week induction phase, followed by monthly injections in the maintenance phase, until disease progression or death.

The primary objectives are to determine the recommended dose of intrathecal QL1706 in combination with pemetrexed and to assess safety based on the incidence of treatment-related adverse events. Clinical response rate, progression-free survival related to leptomeningeal metastasis, and overall survival are also evaluated. Patients undergo cerebrospinal fluid and blood specimen collection to evaluate potential clinical, molecular, and/or immune predictors of treatment efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed diagnosis of solid tumors; Cerebrospinal fluid cytopathology is positive.
2. Male or female aged between 21 and 75 years; Normal liver and kidney function; WBC≥4000/mm3, Plt≥100000/mm3.
3. No history of severe nervous system disease; No severe dyscrasia.

Exclusion Criteria:

1. Any evidence of nervous system failure, including severe encephalopathy, grade 3 or 4 leukoencephalopathy on imaging, and Glasgow Coma Score less than 11.
2. Any evidence of extensive and lethal progressive systemic diseases without effective treatment.
3. A history of HIV or AIDS, acute or chronic hepatitis B or C infection, previous anti-PD1 therapy-induced pneumonitis, or have ongoing >Grade 2 adverse events of such therapy; or ongoing autoimmune disease that required systemic treatment in the past 2 years.
4. Patients with poor compliance or other reasons that were unsuitable for this study.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-03-17 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
PR2D | From date of treatment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 6 months
  The recommended phase II dose. The dose limiting toxicity was defined as ≥ grade 3 neurological toxicities (e.g., chemical meningitis) or other grade 4 toxicity.
Incidence of treatment-related adverse events | From date of treatment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 6 months.
  The incidence of treatment-related adverse events were measured for determining tolerability and safety. Adverse events (AEs) are evaluated according to the Common Terminology Criteria for Adverse Events (CTCAE). Events of grade 3-5 are defined as moderate and severe adverse events.

OTHER OUTCOMES:
Clinical response rate | From date of treatment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 6 months
  The response assessment in neuro-oncology criteria (RANO) proposal for response criteria of leptomeningeal metastasis was used to assess the clinical response in this study.
Progression-free survival related to leptomeningeal metastasis (LMPFS) | From date of treatment until the date of first documented leptomeningeal metastasis progression or date of death from any cause, whichever came first, assessed up to 6 months
  LMPFS was defined as time from the start of treatment until leptomeningeal metastasis progression or death. The leptomeningeal metastasis progression was determined based on the RANO proposal evaluation criteria which have been established and published on Neuro Oncol.
Overall survival(OS) | From the enrollment of this study until date of death from any cause, whichever came first, or the last follow-up, assessed up to 6 months.
  Overall survival was recorded since the date of patient enrollment. All patients were followed up until death or the end of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Zhenyu Pan, PhD,MD, Principal Investigator — The Affiliated HuizhouHospital, Guangzhou Medical University
Locations (1):
- The Affiliated Huizhou Hospital, Guangzhou Medical University, Huizhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No